CLINICAL TRIAL: NCT06088979
Title: A Multicenter Phase 2b Randomized, Double-Masked, Placebo-Controlled Dose-Ranging Study of TOUR006 in Participants With Thyroid Eye Disease
Brief Title: A Study to Investigate Efficacy and Safety of TOUR006 in Participants 18 to 80 Years of Age With Thyroid Eye Disease
Acronym: spiriTED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tourmaline Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOUR006-T01; U1111-1308-4718 (Other: WHO Universal Trial Number (UTN)); 2024-514801-69-00 (Other: EU CTN)
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
Keywords: TED; Graves' Disease; Thyroid Eye Disease; Exophthalmos; Eye Diseases; Thyroid Diseases; Graves' Ophthalmopathy; Hyperthyroidism
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Exophthalmos; Eye Diseases; Thyroid Diseases; Hyperthyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TOUR006 - 20 MG (Experimental): In part A of the study, participants will receive a total of three 20 mg subcutaneous injections: 1 injection every 8 weeks (Day 1, Week 8, Week 16) followed by treatment in part B of the study based on proptosis response and rescue therapy use.
  Interventions: Drug: TOUR006 - 20 MG
- TOUR006 - 50 MG (Experimental): In part A of the study, participants will receive a total of three 50 mg subcutaneous injections: 1 injection every 8 weeks (Day 1, Week 8, Week 16) followed by treatment in part B of the study based on proptosis response and rescue therapy use.
  Interventions: Drug: TOUR006 - 50 MG
- Placebo (Placebo Comparator): In part A of the study, participants will receive a total of three Placebo subcutaneous injections: 1 injection every 8 weeks (Day 1, Week 8, Week 16) followed by treatment in part B of the study based on proptosis response and rescue therapy use.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TOUR006 - 20 MG — TOUR006 20 MG
  Arms: TOUR006 - 20 MG
Other: Placebo — Placebo
  Arms: Placebo
Drug: TOUR006 - 50 MG — TOUR006 - 50 MG
  Arms: TOUR006 - 50 MG

SUMMARY:
Phase 2b trial of TOUR006 in Thyroid Eye Disease (TED) to evaluate 20mg and 50mg doses against placebo given by a subcutaneous injection every eight weeks to TED patients who are in the active inflammatory phase of disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves' disease associated with moderate to severe active TED
* Onset of active TED symptoms within approximately 15 months
* Proptosis (exophthalmos) ≥3 mm above the normal range per investigator judgment (based upon race and gender) for the study eye
* CAS ≥4 (on the 7-item scale) for the study eye
* Presence of TSI >130% of the normal reference standard or >0.55 IU/L (depending on assay method) and laboratory reference ranges

Additional inclusion criteria are defined in the study protocol.

Exclusion Criteria:

* Anticipated need for intervention due to sight-threatening complications or other significant and acute deterioration in vision
* Any previous treatment with teprotumumab or other agent that inhibits the IGF-1 receptor
* History of systemic (eg, oral or IV) steroid use with a cumulative dose equivalent to >1 g of methylprednisolone for the treatment of TED. Previous oral steroid use with a cumulative dose of ≤1g methylprednisolone (or equivalent dosage for other systemic corticosteroid) for the treatment of TED, however, is allowed if the corticosteroid was discontinued at least 6 weeks before baseline (Day 1) and completely tapered by Baseline (if applicable).
* Systemic (oral or IV) corticosteroid use for conditions other than TED within 6 weeks of baseline (Day 1) or not completely tapered by baseline (if applicable).
* Any major illness/condition or evidence of an unstable clinical condition that, in the investigator's judgment, will substantially increase the risk to the participant, or confound the interpretation of safety assessments, if they were to participate in the study
* Any other condition that, in the opinion of the investigator, would impair the ability of the participant to comply with the study procedures or impair the ability to interpret data from the participant's participation in the study
* Pregnant or lactating

Additional exclusion criteria are defined in the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving a proptosis response defined as a ≥2 mm reduction in proptosis from baseline in the study eye without deterioration [≥2 mm increase] of proptosis in the fellow eye and without need for rescue therapy/intervention). | 20 weeks

SECONDARY OUTCOMES:
Percentage of participants achieving a proptosis response with 20mg TOUR006 administered SC every 8 weeks or 50mg TOUR006 administered SC every 8 weeks. | 72 weeks
Percentage of participants attaining a complete or near complete response on the 7-point Clinical Activity Score (CAS). | 72 weeks
Percentage of participants attaining ≥1 grade decrease in diplopia. | 72 weeks
Incidence of Treatment Emergent Adverse Events by severity and Serious Adverse Events through Week 72. | 72 weeks
Mean change from baseline in serum trough concentration of TOUR006. | 72 weeks
Mean change from baseline in serum TSI. | 72 weeks
Percentage of participants with anti-drug antibodies. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Tourmaline Bio
Locations (56):
- United States (30):
  - Catalina Eye Care - Site 840-121, Tucson, Arizona
  - Headlands Research - AMCR - Site 840-131, Escondido, California
  - Foothill Eye Institute - Site 840-116, Pasadena, California
  - University of California Davis Eye Center - Site 840-119, Sacramento, California
  - Cockerham Eye Consultants - Site 840-114, San Diego, California
  - The Pacific Center for Oculofacial and Aesthetic Plastic Surgery - Site 840-122, San Francisco, California
  - UC Hospital Sue Anschulz-Rodgers Eye Center - Site 840-101, Aurora, Colorado
  - Bascom Palmer Eye Institute - Site 840-115, Miami, Florida
  - Cordova Research Institute - Site 840-103, Miami, Florida
  - Aran Eye Associate, Sweetwater, Florida
  - University of Louisville Health Eye Institute - Site 840-108, Louisville, Kentucky
  - Ophthalmic Consultants of Boston - Site 840-128, Boston, Massachusetts
  - W.K. Kellogg Eye Center - Site 840-126, Ann Arbor, Michigan
  - Michigan State University - Site 840-127, East Lansing, Michigan
  - Kahana Oculoplastic and Orbital Surgery - Site 840-112, Livonia, Michigan
  - Mayo Clinic - Site 840-102, Rochester, Minnesota
  - University of Missouri-Kansas City School of Medicine - Site 840-130, Kansas City, Missouri
  - Ophthalmic Plastic, Reconstructive, Orbital & Cosmetic Surgery - Site 840-123, Las Vegas, Nevada
  - Hackensack University Medical Center - Site 840-105, Hackensack, New Jersey
  - Columbia University - Site 840-125, New York, New York
  - University of North Carolina at Chapel Hill - Site 840-104, Chapel Hill, North Carolina
  - Bergstrom Eye Research - Site 840-134, Fargo, North Dakota
  - Eye Physicians, LLC - Site 840-118, Columbus, Ohio
  - Headlands Research - TMA - Site 840-132, Myrtle Beach, South Carolina
  - Academy of Diabetes, Thyroid, and Endocrine - Site 840-129, El Paso, Texas
  - DCT Fort Worth Research Center - Site 840-133, Fort Worth, Texas
  - Neuro-Eye Clinical Trials, Inc - Site 840-106, Houston, Texas
  - Houston Methodist Hospital - Site 840-124, Houston, Texas
  - Sun Research Institute - Site 840-120, San Antonio, Texas
  - University of West Virginia - Site 840-113, Morgantown, West Virginia
- Brazil (8):
  - Freire Pesquisa Clinica - Site 076-773, Belo Horizonte
  - UFG - Hospital de Clinicas da Universidade Federal de Goias - Site 076-762, Goiânia
  - Santa Casa de Misericordia de Porto Alegre - Site 076-767, Porto Alegre
  - Universidade Federal do Rio Grande do Sul (UFRGS) - Site 076-775, Porto Alegre
  - NPCRS - Nucleo de Pesquisa Clinica do Rio Grande do Sul - Site 076-764, Porto Alegre
  - Centro Brasileiro de Pesquisa Clínica - Rio de Janeiro Ltd - Site 076-765, Rio de Janeiro
  - Irmandade da Santa Casa de Misericordia de Sao Paulo - Site 076-771, São Paulo
  - IPEPO - Instituto Paulista de Estudos e Pesquisas em Oftalmologia - Site 076-761, São Paulo
- Canada (2):
  - Ottawa Hospital Research Institute - Site 124-202, Ottawa, Ontario
  - McGill University Health Center - Site 124-201, Montreal, Quebec
- France (2):
  - CHU Angers - Site 250-252, Angers
  - CHU de Nantes - Hopital Nord Laennec - Site 250-251, Nantes
- Italy (3):
  - Azienda Ospedaliera Universitaria Federico II - Site 380-382, Napoli
  - Azienda Ospedaliera Universitaria Federico II - Site 390-382, Napoli
  - Azienda Ospedaliero Universitaria Pisana - Site 380-381, Pisa
- Al-Essra Hospital - Site 400-401, Amman, Jordan
- Latvia (2):
  - Riga East Clinical University Hospital, Clinic Bikernieki - Site 428-901, Riga
  - Ziemelkurzemes Regional Hospital - Site 428-902, Ventspils
- Southern Eye Specialists Ltd - Site 554-501, Christchurch, New Zealand
- University of Puerto Rico, Medical Sciences Campus - Site 630-602, San Juan, Puerto Rico
- Univerzitna nemocnica Bratislava - Nemocnica sv. Cyrila a Metoda - Site 703-211, Bratislava, Slovakia
- South Korea (2):
  - Seoul National University Hospital - Site 410-002, Seoul
  - Seoul St. Mary's Hospital Site 410-001, Seoul
- Spain (3):
  - Hospital La Arruzafa - Site 724-802, Córdoba
  - Hospital Universitario Ramon y Cajal - Site 724-803, Madrid
  - Hospital Universitario Virgen Macarena - Site 724-801, Seville

IPD SHARING:
Plan to Share IPD: No